CLINICAL TRIAL: NCT01373697
Title: Clinical Multicenter, Phase III, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Ibuprofen 50mg/g Gel in the Treatment of Patients With Muscle Pain, Joint, or Pain Caused by Sprains, Contusions, Tendinitis, or Myofascial Compared to Profenid ® 25mg/g. Gel
Brief Title: Study to Assess the Efficacy and Safety of Ibuprofen 50 mg/g Gel Compared to Profenid 25mg/g Gel
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratório Teuto Brasileiro S/A (Industry)
Responsible Party: PHC Pharma Consulting, Dagoberto Brandão
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEU-IBU- 01-10
Record Dates: First submitted 2011-03-22; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Muscular Atrophy; Sprains; Tendonitis
Keywords: Ibuprofen; muscle pain; sprains; contusions; tendonitis
MeSH Terms: conditions — Muscular Atrophy; Sprains and Strains; Tendinopathy; Myalgia; Contusions | interventions — Ibuprofen; Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Profenid (Active Comparator): Apply the gel on the spot of pain or injury, massaging slightly to facilitate the penetration of 8 in 8 hours during 5 days. Leave the gel on the the site at least 4 hours before removal
  Interventions: Drug: Profenid
- Ibuprofen (Active Comparator): Apply the gel on the spot of pain or injury, massaging slightly to facilitate the penetration of 8 in 8 hours during 5 days. Leave the gel on the the site at least 4 hours before removal
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Apply the gel at the site of pain or injury, massaging gently to promote penetration of 8 in 8 hours for 5 days. Leave the gel on the premises at least 4 hours before removal
  Arms: Ibuprofen
Drug: Profenid — Apply the gel on the spot of pain or injury, massaging slightly to facilitate the penetration of 8 in 8 hours during 5 days. Leave the gel on the the site at least 4 hours before removal
  Arms: Profenid

SUMMARY:
The aim of this study is to determine that ibuprofen 50mg/g gel is effective and safety treating patients with muscle aches, joint pains or due to sprains, bruises, tendinitis or myofascial compared to Profenid 25mg/g gel.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the efficacy of ibuprofen 50 mg/g gel in the treatment of patients with muscle, joint pain caused by sprains, contusions, tendinitis, or myofascial compared to Profenid 25mg/g gel.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, of any race, aged 12 years;
* Ability to read, understand and sign the Informed Consent in the case of minors monitoring and consent of a parent;
* Complaint of clinical muscle pain, joint pain caused by sprains, contusions, tendonitis, or myofascial;
* Score more than 4 VAS symptom reviewed: Pain;
* Patients able to understand and follow the protocol of the trial.
* Patients with or without ligament injury ligament injury partial and incomplete

Exclusion Criteria:

* Known hypersensitivity to components of the formula, both the medication and the comparative test;
* Hypersensitivity to acetylsalicylic acid;
* Hypersensitivity to ketoprofen, ibuprofen or other anti-inflammatory steroid;
* Hypersensitivity to acetaminophen;
* Skin changes in the pathological site of application, such as eczema or acne, or infected skin or wound;
* Pregnant or lactating women.
* Patients who require surgery or immobilization;
* Patients with fractures or ligament rupture;
* Patients taking anticoagulants;
* Patients with decompensated concomitant systemic diseases, such as diabetes, congenital or acquired blood disorders, convulsive disorders, autoimmune diseases, renal failure, severe infections, hormonal disorders and pulmonary disorders;
* Use of NSAIDs, corticosteroids or venotherapics, threads or any other form of administration;
* History of alcoholism or substance abuse;
* Conditions in the opinion of the investigator make the patient unsuitable to participate in the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Clinical study evaluating the efficacy and safety of Ibuprofen 50mg / g gel in the treatment of patients with muscle pain, joint, or pain caused by sprains, contusions, tendinitis, or myofascial compared to Profenid ® 25mg / g gel. " | five days
  To evaluate the efficacy of ibuprofen 50 mg / g gel in the treatment of patients with muscle aches, joint pains or due to sprains, bruises, tendinitis or myofascial compared with Profenid® Gel 25mg / g, will be used two methods. 1. the visual analog scale (VAS)and 2. investigator's opinion to measure before and after treatment comparing the decrease of the symptoms. The study will have 144 patients to be included with any sex or race, minimum age 12 years.

SECONDARY OUTCOMES:
Clinical study evaluating the tolerability of Ibuprofen 50mg / g gel in the treatment of patients with muscle pain, joint, or pain caused by sprains, contusions, tendinitis, or myofascial compared to Profenid ® 25mg / g gel. " | five days
  To evaluate the tolerability of ibuprofen 50 mg / g gel in the treatment of patients with muscle aches, joint pains or due to sprains, bruises, tendinitis or myofascial compared with Profenid ® Gel 25mg / g will be use a measure using Naranjo algorithm to determinate the causality of the events.

CONTACTS AND LOCATIONS:
Overall Officials: Abel Pereira, investigator, Principal Investigator — ABC School Medicine
Locations (1):
- ABC School of Medicine, São Paulo, Brazil